CLINICAL TRIAL: NCT05558163
Title: Minimally Invasive Scrotal Incision for Penile Prosthesis Implantation, Novel Technique.
Acronym: PPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Almetwally Algammal,MD, clinical professor, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61158m2
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Penile Prosthesis Infection; Penile Prosthesis; Complications, Infection or Inflammation
Keywords: erectyle dysfunction; penile prothesis
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Intervention Model Description: Patients who will undergo scrotal approach will be compared with a case-matched of patients who underwent PPI through peno-scrotal approach in our institution during the last 5 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PPI through traditional penoscrotal approach (Other): cases of erectyl dysfunction who underwent PPI throug penoscrotal approach
  Interventions: Procedure: penoscrotal approach for PPI
- PPI through novel transverse scrotal approach (Other): cases of erectyl dysfunction who underwent PPI throug novel transverse scrotal approach
  Interventions: Procedure: transverse scrotal approach for PPI

INTERVENTIONS:
Procedure: transverse scrotal approach for PPI — penile prothesis implantation through penoscrotal approach outcome
  Arms: PPI through novel transverse scrotal approach
Procedure: penoscrotal approach for PPI — penile prothesis implantation through penoscrotal approach outcome
  Arms: PPI through traditional penoscrotal approach

SUMMARY:
The main goals of this study are to examine the superiority of this novel technique and its acceptance by patients with ED candidate for PPI and compare these results with data available in the literature for ordinary peno-scrotal incision.

DETAILED DESCRIPTION:
Rational for the expected superiority of scrotal approach over peno-scrotal approach in penile prosthesis implant (PPI):

A- Expected to have all the previously mentioned pros of the traditional approach.

B- Expected lower incidence of post-operative pain with our novel approach owing to lower sensitivity of scrotal skin and tension free wound closure compared to traditional peno-scrotal approach.

C- Expected lower incidence of infection owing to multilevel wound closure done in our novel approach.

D- Expected rapid wound closure and wound healing than traditional peno-scrotal approach owing to difference in embryologic origin of penile and scrotal skin.

E- Validity of this novel approach for malleable and inflatable prosthesis implantation.

F- Short learning curve owing to simplicity of the approach even for junior urologists.

3- Research methodology

- Responsible party: drmohamedalgammal@gmail.com Study Type: Interventional study Sampling: Hospital-based sample Estimated Enrollment: 200 participants Intervention Model: Patients who will undergo scrotal approach will be compared with a case-matched of patients who underwent PPI through peno-scrotal approach in our institution during the last 5 years.

Study Start Date: 2022

Estimated Study Completion Date: 2023

Study Location:

Al-Hussin and Sayed Galal, Al-Azhar University Hospital, Cairo, Egypt.

Study Population:

- The study participants are male patients who are candidate for penile prosthesis implantation and will accept to do minimal scrotal incision procedure for treatment of ED.

Study Sample:

- All available cases with complete medical record and accepted follow-up with us will be included.

Pre-Operative Evaluation

1. Full medical history taking including full sexual history and (IIEF5) table 1.
2. Physical Examination including general, abdominal and local genital examination.
3. Laboratory investigations:

   1. Complete urine analysis and urine culture
   2. Blood chemistry tests include blood urea, serum creatinine, liver function tests, blood sugar, and coagulation profile.
   3. Lipid profile.
   4. Hormonal assessment including serum testosterone, Follicular stimulating hormone (FSH) Luteinizing hormone (LH) and prolactin.
   5. Complete blood cell count (CBC).
   6. Psychosexual assessment if needed.
4. Imaging:

   1. Penile douplex Ultra-sonography.
   2. Nocturnal penile tumescence and rigidity study, (NPTR or Rigiscan) if needed.
   3. Abdomino-pelvic ultra-sonography with residual urine calculation.
   4. Uroflowmetry if needed.
5. Cardiopulmonary assessment

Post-operative evaluation:

* Post-operative CBC.
* Post-voiding residual urine volume.
* (Qmax.) maximum flow rate.
* Regular post-operative assessment of

  1. Pain using Numeric Pain Rating Scale (NRS)
  2. Wound healing, cosmetic appearance after healing and any incidence of infection.
  3. Incidence of satisfaction after regaining sexual activity using SSI.

ELIGIBILITY:
Inclusion Criteria:

The study participants are male patients who are candidate for penile prosthesis implantation and will accept to do minimal scrotal incision procedure for treatment of ED.

Exclusion Criteria:

* male patients with active scrotal infection.
* contraindicaions to anasthesia.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective cure rate | 3 to 4 weaks
  will be judged according to rate of wound healing, cosmotic final results, scar tension and scar pain.
Objective cure rate | 4-12 weaks
  should include rate of complications as fistula, scar, extensive fibrosis, infection rate, incidence of prosthetic removal.